CLINICAL TRIAL: NCT04026191
Title: A Prospective, Open-Label, Multi-Center Post-Market Clinical Follow-Up Study to Evaluate the Residual Risk of OrthoVisc®-T (OVT) in the Treatment of Chronic Lateral Epicondylosis (Tennis Elbow)
Brief Title: OVT for Epicondylosis (Tennis Elbow)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVT 16-03
Record Dates: First submitted 2019-07-10; First posted 2019-07-19 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Epicondylitis, Lateral; Tendinopathy, Elbow
Keywords: Hyaluronic Acid; Sodium Hyaluronate
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthovisc-T (Other)
  Interventions: Device: OrthoVisc®-T (OVT)

INTERVENTIONS:
Device: OrthoVisc®-T (OVT) — Sodium hyaluronate supplied as a 2 mL (15mg/mL) unit dose in a 3 mL glass syringe.

SUMMARY:
To assess the residual risk of OrthoVisc-T (OVT) for the treatment of chronic lateral epicondylosis (Tennis Elbow). This trial will provide clinical data on a subject population not previously researched which have failed prior treatments for lateral epicondylosis.

DETAILED DESCRIPTION:
Orthovisc-T is a sterile viscoelastic preparation supplied in a disposable glass syringe containing 2.0 mL of sodium hyaluronate (15 mg/mL) dissolved in physiological saline. The Orthovisc-T device is intended to relieve pain and restore function in tendons affected by chronic lateral epicondylosis. The hyaluronic acid solution provides extracellular supplementation of the elbow with lateral epicondylosis, lubricating and hydrating the affected site, thereby providing the ideal environment for healing of the damaged tissue.

The objective of the study is to evaluate the residual risk of two peri-osteotendinous injections of Orthovisc-T spaced one week apart for the relief of elbow pain and to restore function in patients with lateral epicondylosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of chronic lateral epicondylosis defined as:

   1. Pain reproducible on palpation of the lateral epicondyle / common extensor origin, and
   2. Pain reproducible during resisted wrist extension
3. Failed prior treatment for lateral epicondylosis
4. Able and willing to provide signed informed consent.
5. Subject must be willing to abstain from other peri-articular treatments of the elbow for the duration of the study.
6. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
7. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol.

Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan
2. Infection or skin disease in the area of the injection site or elbow joint
3. Subject received a peri-articular injection of Hyaluronic Acid (HA) and/or steroid in either elbow within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either elbow during the course of this study.
4. Known inflammatory or autoimmune disorders, or other pre-existing medical conditions that, in the opinion of the investigator, could impact healing or affect the ability of the subject to complete the study and comply with the study requirements.
5. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
6. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index elbow only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index elbow is allowed.
7. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
8. Subject was involved in any other research study involving an investigational product, or a new application of an approved product, within 60 days of signing the ICF.
9. Subject is receiving or in litigation for worker's compensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The mean change in Elbow Pain from Baseline to 6 Months | From baseline to 6 months
  The mean change in Pain After Grip from Baseline to 6 Months as measured with a 0-10 Likert Scale comparing the OVT group to Baseline measurements.

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - FN Motol (University Hospital Motol) Klinika dětské a dospělé ortopedie a traumatologie 2.LF UK a FN v Motole, Prague
  - MEDICAL Plus, Uherské Hradiště
  - "Krajská zdravotní Masarykova nemocnice, Ústí nad Labem Ortopedické oddělení", Ústí nad Labem

IPD SHARING:
Plan to Share IPD: No